CLINICAL TRIAL: NCT03182075
Title: Emotional Reactivity Training for Obsessive-Compulsive and Related Disorders
Brief Title: Computerized Training for Individuals Diagnosed With Obsessive-Compulsive and Related Disorders
Acronym: EmRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 40185
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; OCD; Obsessive Personality Disorder; Compulsive Behavior; Personality Disorders; Mental Disorders; Anxiety Disorders; Impulsive Behavior; Cognition; Emotion; Emotional Regulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Compulsive Personality Disorder; Compulsive Behavior; Personality Disorders; Mental Disorders; Anxiety Disorders; Impulsive Behavior; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Training (Experimental): OCD and hoarding disorder participants will receive active emotional reactivity training (14 sessions) via computer.
  Interventions: Behavioral: Computerized Training
- Passive Training (Sham Comparator): OCD and hoarding disorder participants will receive passive computerized training (14 sessions) via computer.
  Interventions: Behavioral: Computerized Training

INTERVENTIONS:
Behavioral: Computerized Training — OCD and hoarding disorder participants will receive 14 sessions of training via computer within 3 weeks.

SUMMARY:
Obsessive-Compulsive Disorder (OCD) is a chronic and disabling disorder that costs the economy over $2 billion annually and represents a significant public health problem. This study aims to build on our understanding of aberrant emotional processing in OCD. The proposed project tests whether a computerized training aimed to alter emotional processes, can relieve repetitive thoughts and behaviors.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years old and older
* primary diagnosis of OCD
* sufficient severity of OCD symptoms
* Stable on psychotropic or other medication
* capacity to provide informed consent

Exclusion criteria:

* psychiatric or medical conditions that make participation unsafe
* concurrent use of any medications that might increase the risk of participation
* concurrent Cognitive-Behavioral therapy for OCD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (for participants diagnosed with OCD) | up to 2 months
  Improvement in OCD severity is measured by the YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response is defined as at least a 35% reduction on the YBOCS.
Savings Inventory Revised Scale (for participants diagnosed with hoarding disorder) | up to 2 months
  The SI-R is a 23-item questionnaire with 3 factor-analytically defined sub-scales for difficulty discarding, excessive clutter, and compulsive acquisition.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Rodriguez Lab Website — http://rodriguezlab.stanford.edu